CLINICAL TRIAL: NCT06708754
Title: PBM-LEF Study: The Impact of PBM on Biomarkers of Radiation Lymphedema and Fibrosis in Head and Neck Cancer Patients: A Feasibility Study
Brief Title: Impact of Photobiomodulation (PBM) on Biomarkers of Radiation Lymphedema and Fibrosis in Head and Neck Cancer Patients
Acronym: PBM-LEF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-00511
Record Dates: First submitted 2024-11-26; First posted 2024-11-27 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Radiation Lymphedema; Radiation Fibrosis; Head and Neck Cancer
MeSH Terms: conditions — Radiation Fibrosis Syndrome; Head and Neck Neoplasms | interventions — Low-Level Light Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Treatment: PBM Therapy (Experimental): Participants who received bilateral neck RT will be treated with PBM to a total of 12 sites - 6 sites on each side of the neck and face along the 3 neck nodal levels (II, III, IV) of the sternocleidomastoid muscle (SCM), along the major salivary glands (parotid, and submandibular) and masseter].
  Treatment will occur at two timepoints:
  * At least 3 months and less than 18 months after RT completion of last dose to any site
  * Between 18 and 36 months after RT completion of last dose to any site
  Interventions: Device: Photobiomodulation (PBM) Therapy
- Sham Treatment (Sham Comparator): Participants who received bilateral neck RT will be treated with SHAM PBM to a total of 12 sites - 6 sites on each side of the neck and face along the 3 neck nodal levels (II, III, IV) of the sternocleidomastoid muscle (SCM), along the major salivary glands (parotid, and submandibular) and masseter].
  Treatment will occur at two timepoints:
  * At least 3 months and less than 18 months after RT completion of last dose to any site
  * Between 18 and 36 months after RT completion of last dose to any site
  Interventions: Device: Sham PBM

INTERVENTIONS:
Device: Photobiomodulation (PBM) Therapy — PBM is a low-intensity form of light therapy and employs visible or near-infrared (NIR) light generated from a laser or Light Emitting Diode (LED).
  In this study, PBM will be delivered using an LED device emitting 660 and 850nm with the purpose of research. The output power typically ranges from 5 to 200 mW with wavelengths ranging 600-1,000nm.
  Arms: Active Treatment: PBM Therapy
Device: Sham PBM — Sham PBM will be delivered using a matching shame device that emits no output power.
  Arms: Sham Treatment

SUMMARY:
Radiation fibrosis syndrome (RFS) is a general side effect of radiation therapy (RT) which can adversely impact patients chronically over years typically triggered by an acute inflammatory state that evolves into chronic inflammation and tissue remodeling causing lymphedema, fibrosis, pain, atrophy and organ dysfunction. Some of the side effects that encompass RFS in the head and neck (HNC) population include decreased ability to fully open the mouth (trismus), neck pain and tightness (cervical dystonia), lymphedema (swelling), difficult with speech and swallowing and salivary hypofunction. Although there is Level I evidence demonstrating the benefit of Photobiomodulation (PBM) therapy to prevent acute mucositis in HNC patients treated with RT, there is only limited data regarding its impact.

This is a clinical trial to compare active treatment (PBM-therapy) with sham control (Sham- therapy). Up to 60 patients will be randomized to the two groups with equal allocation to estimate the efficacy (soft tissue thickness) of external Photobiomodulation (PBM) with light-emitting diode (LED) planned therapy for the treatment of radiation fibrosis syndrome (RFS) in head and neck cancer (HNC) patients who have undergone radiation therapy (RT) compared with sham control.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with radiation for head and neck cancer who are ≥ 3 months < 36 months post-RT (last RT).
* Patients who received at least 50Gy of bilateral neck RT. Subjects who received RT or concurrent chemoradiation (chemoRT) therapy for HNC are eligible.
* No evidence of disease as documented by imaging 3 months after completion of RT.
* Common Terminology Criteria for Adverse Events (CTCAE) fibrosis score ≥ 2 at enrollment.
* Patient who has body mass index (BMI) >30 at the time of enrollment may be excluded at a discretion of the principal investigator if fibrotic areas cannot be identified by clinical objective assessment of fibrosis.
* Willing to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* Woman who are pregnant or planning to become pregnant or breast-feeding.
* Patients enrolled on another drug or device investigational trial for prevention or treatment of LEF.
* Patients deprived of freedom, under supervision or guardianship.
* Patients unable to attend to scheduled visits due to geographical, social or mental reasons.
* Patients who received prior PBM therapy for RT toxicities in the last year;
* Patients who report being photosensitive.
* Patients who have chronic immunosuppression or are on current immunosuppressive therapies.
* Any patient who, in the opinion of the investigator, is unable or unlikely to comply fully with the study requirements or procedures for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Soft tissue thickness (STT) at Nodal Level II - Right Side | Baseline, Week 2 Post-Treatment
  STT will be measured via ultrasound.
STT at Nodal Level II - Left Side | Baseline, Week 2 Post-Treatment
  STT will be measured via ultrasound.
STT at Nodal Level III - Right Side | Baseline, Week 2 Post-Treatment
  STT will be measured via ultrasound.
STT at Nodal Level III - Left Side | Baseline, Week 2 Post-Treatment
  STT will be measured via ultrasound.
STT at Nodal Level IV - Right Side | Baseline, Week 2 Post-Treatment
  STT will be measured via ultrasound.
STT at Nodal Level IV - Left Side | Baseline, Week 2 Post-Treatment
  STT will be measured via ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Hu, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States